CLINICAL TRIAL: NCT05315869
Title: Retrocaecal Appendicitis: Risk Factor for Perioperative Complications?
Brief Title: a Retrospective Observational Study Comparing Outcomes of Retrocaecal Appendicitis With Non-retrocaecal Appendicitis
Status: Completed | Type: Observational
Sponsor: Faculty Hospital Kralovske Vinohrady (Other Government)
Responsible Party: Principal Investigator, Adam Whitley, MUDr., Faculty Hospital Kralovske Vinohrady
Other Study IDs: AppendicitisFNKV
Record Dates: First submitted 2022-03-20; First posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Appendicitis; Appendicitis Acute; Retrocecal Appendicitis
MeSH Terms: conditions — Appendicitis | interventions — Appendectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrocaecal group: Patients who underwent surgery for signs of acute appendicitis and had intraoperative finding of the appendix located in the retrocaecal position.
  Interventions: Procedure: Appendectomy
- Non-retrocaecal group: Patients who underwent surgery for signs of acute appendicitis and had intraoperative finding of the appendix not located in the retrocaecal position.
  Interventions: Procedure: Appendectomy

INTERVENTIONS:
Procedure: Appendectomy — Surgical procedure for removal of the appendix

SUMMARY:
A retrospective observational study investigating whether retrocecal appendicitis associated with worse operative and postoperative outcomes than non-retrocecal appendicitis.

DETAILED DESCRIPTION:
Acute appendicitis is the most common cause of acute abdomen requiring acute surgery. The prevalence of the retrocaecal position of the appendix varies significantly between studies from 14 to 36%. Appendectomy of a retrocecal appendix is generally considered to be more demanding procedure than appendectomy of appendices in other positions. The aim of this study is to investigate whether retrocaecal appendicitis is associated with a higher rate of perioperative complications and delayed diagnosis when compared with the other positions.

A retrospective analysis of prospectively collected data of patients undergoing surgery for signs of acute appendicitis from January 2015 to April 2020 at the University Hospital Kralovske Vinohrady. Two groups of patients were be formed: the retrocaecal group and the non-retrocaecal group.

The following data were recorded: sex, age, body mass index, length of hospital stay, abdominal drain placement, length of surgery, surgical approach (laparoscopic, open or converted), operative finding (normal appendix or catarrhal, phlegmonous, gangrenous, or perforated appendicitis), position of the appendix (retrocaecal or non-retrocaecal positions), histopathological findings (acute inflammation, chronic inflammation, appendiceal tumour or normal appendix), 30-day postoperative complications, 30-day postoperative mortality, symptoms (abdominal pain, nausea, vomiting, diarrhoea, body temperature above 37 degrees celsius, urological complaints and gynaecological complaints), duration of symptoms (from onset to surgery), serious comorbidities and diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing surgery for signs of acute appendicitis at the department of surgery of the University Hospital Kralovske Vinohrady between January 2015 to April 2020

Exclusion Criteria:

* Patients under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients of the treated at the department of surgery of the University Hospital Kralovske Vinohrady
Sampling Method: Non-Probability Sample
Enrollment: 754 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Number of patient with postoperative complications | 30 days after intervention (appendectomy)
  surgical site infections, postoperative ileus, bleeding, internal complications,
Number of patient who undergo converted appendectomy | during the surgery
  Conversion from laparoscopic to open appendectomy
Length of hospital stay | 30 days after intervention (appendectomy)
  Length of hospital stay after the procedure in days
Duration of procedure | Throughout the study period (1/2015-4/2020)
  Duration of appendectomy in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Adam Whitley, MUDr., Study Chair — University Hospital Kralovske Vinohrady
Locations (1):
- Adam Whitley, Prague, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No